CLINICAL TRIAL: NCT03456687
Title: Effects of Exenatide on Motor Function and the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201703187 - N; R01NS052318 (NIH); OCR17539 (Other: Universiy of Florida)
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Parkinson's Disease
Keywords: Exenatide
MeSH Terms: conditions — Parkinson Disease | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exenatide (Experimental): This group will receive a weekly Exenatide 2mg injection for one year.
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Exenatide will be administered through a subcutaneous injection once per week for the duration of the study (1 year).
  Other Names: Bydureon; Glucagon-like peptide-1 receptor agonist

SUMMARY:
The purpose of this research study is to investigate how the brain and motor behavior changes Parkinson's Disease (PD) over time in response to Exenatide. In previous clinical trials, PD patients have experienced symptomatic improvement on Exenatide and literature suggests it may help slow the progression of Parkinson's. Both will be evaluated in this study.

DETAILED DESCRIPTION:
Participants will receive baseline testing to confirm a diagnosis of Parkinson's Disease and to determine eligibility in the research study. All of the participants in this study will receive the study drug (Exenatide). The study drug will be provided at the end of the first visit, and participants will be administered the drug once per week for the duration of the study (1 year).

During the research study the following test may occur: (1) questionnaires about quality of life and depression; (2) tests to measure strength and motor function; (3) tests to measure cognition; (4) orientation session to learn a precision gripping task; (5) functional MRI scan of the brain; (6) structural MRI scan of the brain.

ELIGIBILITY:
Inclusion Criteria:

* patients clinically diagnosed with Parkinson's disease (PD) through use of the UK PD brain bank diagnostic criteria
* early stage PD patients within 5 years of diagnosis who have never taken Exenatide for any reason
* PD patients with a Hoehn and Yahr stage less than or equal to 2 when on medication
* patients able and willing to sign informed consent.

Exclusion Criteria:

* individuals who have any type of implanted electrical device (such as a cardiac pacemaker or a neurostimulator)
* individuals with a certain type of metallic clip in the body (i.e., an aneurysm clip in the brain)
* claustrophobia
* women who are or might be pregnant and nursing mothers. Pregnancy tests will be carried out for each female subject prior to the MRI scan.
* psychiatric disorders or dementia
* other neurologic and orthopedic problems that impair hand movements and walking
* individuals actively participating in another trial of a device, drug or surgical treatment for Parkinson's disease
* individuals who have a history metalworking involving cutting processes such as grinding, filing, shaving, and threading, will need radiological clearance to participate in this study. Specifically, individuals who report a history of metalworking will be referred to Radiology at Shands University of Florida(UF) for an orbitofrontal x-ray.
* individuals who have sustained an eye injury involving metal will also be referred to Radiology at Shands UF for an orbitofrontal x-ray.
* prior stroke or brain tumor
* cognitive impairment as assessed by a Montreal Cognitive Assessment score < 23
* individuals unwilling to comply with the study procedures
* history of gallstones, digestion problems (such as gastroparesis), severe gastrointestinal disease, history of pancreatitis, a thyroid tumor or cancer, pancreas tumor, or kidney problems
* severely impaired renal function with creatinine clearance less than 30 ml/min
* hyperlipidemia defined as more than two times the upper limit of normal
* body mass index less than 18.5
* previous exposure to Exenatide
* diabetes

Ages: 40 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Change in free-water accumulation in the substantia nigra | Baseline and one-year
  12-month study in PD to watch the effect of Exenatide on the progressive increase of free-water accumulation in the substantia nigra.
Change in blood oxygen level-dependent(BOLD) signal in the posterior putamen. | Baseline and one-year
  12-month study in PD to watch the effect of Exenatide on BOLD signal in the posterior putamen.
Change in blood oxygen level-dependent(BOLD) signal in M1. | Baseline and one-year
  12-month study in PD to watch the effect of Exenatide on BOLD signal in M1.
Change in blood oxygen level-dependent(BOLD) signal in the supplementary motor area(SMA). | Baseline and one-year
  12-month study in PD to watch the effect of Exenatide on BOLD signal in the SMA.

CONTACTS AND LOCATIONS:
Overall Officials: David Vaillancourt, PhD, Principal Investigator — University of Florida
Locations (1):
- Laboratory for Rehabilitation Neuroscience, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No